CLINICAL TRIAL: NCT04023370
Title: Evaluation of the Efficacy and Safety of the Application of BeGraft Peripheral Stent Graft System in Interventional Treatment of Revascularisation for Primary Iliac Artery Stenosis and/or Occlusive Lesions: a Prospective, Multi-centre, Randomised Controlled Clinical Study
Brief Title: Evaluation of the Efficacy and Safety of the Application of BeGraft Peripheral Stent Graft System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bentley InnoMed GmbH (Industry)
Collaborators: Shanghai Micro Medical Devices Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT02-01 BGP-China
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Iliac Artery Stenosis

STUDY DESIGN:
Intervention Model Description: Prospective, multi-centre, randomised controlled trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BeGraft Peripheral Stent Graft System (Experimental): Covered stent
  Interventions: Device: Treatment of primary iliac artery stenosis and/or occlusive lesions
- Bare metal stent system (Active Comparator): bare metal stent
  Interventions: Device: Treatment of primary iliac artery stenosis and/or occlusive lesions

INTERVENTIONS:
Device: Treatment of primary iliac artery stenosis and/or occlusive lesions — Stent implantation

SUMMARY:
The trial will be conducted to evaluate the safety and efficacy of the BeGraft Peripheral Stent Graft System in interventional revascularisation for subjects with primary iliac artery stenosis and/or occlusive lesions by conducting a multi-centre, randomised controlled clinical study with a bare metal stent system as the control, thus providing a basis for the formal use of the product in China

DETAILED DESCRIPTION:
This study adopts a prospective, multi-centre, randomised controlled trial design, aiming at evaluating the efficacy and safety of the BeGraft Peripheral Stent Graft System for primary iliac artery stenosis and/or occlusive lesions. A total of 182 subjects are planned to be enrolled, with all consecutively enrolled subjects being randomly assigned to an experimental group (BeGraft group, n=91) and a control group (bare metal stent group, n=91) in the ratio of 1:1 and respectively treated using the BeGraft Peripheral Stent Graft System and the bare metal stent system. Follow-up visits are carried out for the above-mentioned 182 subjects at baseline, upon discharge from hospital, at 30 days, 6 months, 12 months and then once a year from the 2nd to 5th year following surgery. A Doppler ultrasound (DUS) examination is carried out when subjects return to hospital at 6 months following surgery, and a CT angiography (CTA) examination when returning 12 months following surgery, with telephone follow-ups being conducted at 30 days and then once a year from the 2nd to 5th year following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old, no restrictions in terms of male or female;
* Participating in the trial voluntarily, and having signed the informed consent form;
* TASC class A, B, C or D lesions of the common iliac artery and/or external iliac artery;
* Primary iliac atherosclerotic stenosis and/or occlusive lesions;
* Total length of lesions on the affected side ≤100 mm.

Exclusion Criteria:

* Expected survival period <12 months;
* Pregnant women or those unable to take effective contraceptive measures during the trial;
* Aneurysms present close to the target lesion;
* Acute or subacute thrombosis within the target vessel;
* Previously unobstructed internal iliac artery being blocked (diameter stenosis <70%) by the stented region;
* Total occlusive lesions, with the guidewire being unable to return the true lumen in the iliac artery;
* Severe calcification at the target lesion, with the catheter being unable to pass;
* Allergic to cobalt-chromium alloy (L605), ePFTE coating material, carbon coating, contrast agent, antiplatelet agents, anticoagulant drugs or presenting with contraindications;
* Total occlusion of the superficial femoral artery and deep femoral artery, with there being no outflow tract;
* Suffering from extensive diffuse disease at the distal end, resulting in poor blood flow in the outflow tract following stent placement;
* A history of coagulation disorders;
* The subject's mental state making it impossible for them to comprehend the nature, extent and possible consequences of the trial, or having a language barrier making it difficult for the subject to give their informed consent;
* Poor cooperation or potentially poor compliance with the protocol which may cause deviations during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate | 12 month
  The primary patency rate is defined as the absence of restenosis in the treated vessel segment without accompanying target lesion revascularisation (TLR) or amputation.

SECONDARY OUTCOMES:
Device/Surgical success rate | 30 days, 6 months and 12 months following surgery, and then once a year from the 2nd to 5th year following surgery
  Stent placement and integrity

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Beijing Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Shanghai Ninth People's Hospital, Shanghai
  - Suzhou Municipal Hospital, Suzhou
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - General Hospital of Tianjin Medical University, Tianjin
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Tianjin First Center Hospital, Tianjin
  - The Central Hospital of Wuhan, Wuhan
  - The First Hospital of Zhejiang Province, Zhejiang

IPD SHARING:
Plan to Share IPD: No